CLINICAL TRIAL: NCT05147051
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of REAMBERIN® (Meglumine Sodium Succinate) Used for Correction of Metabolic Acidosis in Critically Ill Patients
Brief Title: Meglimine Sodium Succinate for Correction of Metabolic Acidosis in Critically Ill Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Collaborators: Atlant Clinical Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RB-II-2020
Record Dates: First submitted 2021-10-22; First posted 2021-12-07 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Metabolic Acidosis
Keywords: metabolic acidosis; critical illness; acid-base disorder
MeSH Terms: conditions — Acidosis; Critical Illness | interventions — Reamberin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reamberin group (Experimental): Patients receive the investigational treatment (meglumine sodium succinate), 500 ml intravenously every 8 hours (up to 6 infusions).
  Interventions: Drug: Meglumine Sodium Succinate
- Placebo (Placebo Comparator): Patients receive a Placebo (Ringer's solution), 500 ml intravenously every 8 hours (up to 6 infusions).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meglumine Sodium Succinate — 500 ml of 1.4% solution IV at a rate of at least 4 ml and not more than 10 ml per minute
  Arms: Reamberin group
Drug: Placebo — Ringer's solution, 500 ml IV at a rate of at least 4 ml and not more than 10 ml per minute
  Arms: Placebo

SUMMARY:
An acid-base imbalance, called metabolic acidosis (acid-base disorder lasting from several minutes to several days, caused by a decrease in serum bicarbonate ion (HCO3) concentration), is often observed in critically ill patients with various underlying diseases. Metabolic acidosis has a negative impact on the cardiovascular, respiratory, digestive, nervous, excretory, hematological, endocrine, musculoskeletal and immune systems and is associated with unfavourable outcomes. Reamberin® is a solution of disubstituted sodium salt of succinic acid, which has an alkaline reaction and succinate is capable to integrate into the Krebs cycle and restore energy metabolism in the cell. The aim of the present study is to evaluate the efficacy and safety of meglumine sodium succinate at a dose of 500 to 3000 ml in critically ill patients with metabolic acidosis and choose the optimal volume of its solution for the correction of metabolic acidosis in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Informed Consent (if unconscious due to a critical condition, the decision is made by a Council consisting of 3 physicians)
2. Male and female patients aged 18-70
3. Critical illness ((shock (including traumatic, hypovolemic), major trauma, acute massive blood loss, acute complicated surgical diseases of the abdominal organs) accompanied by metabolic acidosis, defined as serum bicarbonate <22mmol/L
4. pH of arterial blood 7.20-7.35, inclusive
5. Planned volume of infusion >= 1500 ml per day
6. Interval between admission to the ICU and randomization <24 hours

Exclusion Criteria:

1. Pregnant and lactating women
2. Known hypersensitivity to any component of the study drug / placebo
3. Chronic kidney disease stage C5 (end-stage renal failure)
4. Acute hepatic failure (ALT > 15 upper normal limits) or liver cirrhosis
5. Traumatic brain injury accompanied by cerebral edema
6. Previously diagnosed mental illness
7. Any chronic disease in the terminal stage with a life expectancy of < 3 months
8. HIV infection
9. Clinically significant cardiovascular disease (unstable angina pectoris or angina pectoris of functional class III or higher; chronic heart failure III - IV class according to NYHA; acute myocardial infarction within 6 months before screening)
10. Extremely low or extremely high body fat
11. Infusion sodium bicarbonate, sodium bicarbonate, trometamol, Sterofundin, Quintasol, Ringer's lactate (Hartmann's solution) within 6 hours before screening
12. Acute respiratory acidosis
13. Poisoning with chemical compounds causing metabolic acidosis
14. Alcohol in saliva at screening >= 0.5 pro mille
15. Previously diagnosed chronic obstructive pulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Elimination of acidosis at 24 hours after the start of treatment | 24 hours
  The proportion of patients who have achieved normalization of the serum bicarbonate level (normalization = serum hydrocarbonate ion concentration ≥22 mmol / Liter), at 24 hours after the start of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Yu Kirov, Principal Investigator — GBUZ Arkhangelsk region "First GKB named after E.E. Volosevich"
Locations (6):
- Russia (6):
  - GBUZ Arkhangelsk region "First GKB named after E.E. Volosevich", Arkhangelsk
  - Ivanovo Regional Clinical Hospital, Ivanovo
  - Central Clinical Hospital with a polyclinic of the Office of the President of the Russian Federation, Moscow
  - Privolzhsky District Medical Center, Nizhny Novgorod
  - Saint-Petersburg I.I.Dzanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - National Research Mordovian State University n.a. N.P. Ogarev, Saransk

IPD SHARING:
Plan to Share IPD: No